CLINICAL TRIAL: NCT04609462
Title: A Trial of High-Flow Nasal Cannula vs. Conventional Oxygen Therapy in Patients With SARS-CoV-2-Related Acute Respiratory Failure: the HiFlo-COVID Trial.
Brief Title: High-Flow Nasal Cannula in Severe COVID-19 With Acute Hypoxemic Respiratory Failure.
Acronym: HiFlo-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001635
Record Dates: First submitted 2020-09-24; First posted 2020-10-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Acute Hypoxemic Respiratory Failure
Keywords: Acute Hypoxemic Respiratory Failure; SARS-CoV-2 infection; High flow nasal cannula; Conventional oxygen therapy; Oxygen therapy
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Phase II, multicenter, randomized, open-label, controlled study of the use of high flow nasal cannula respiratory support vs. conventional oxygen therapy in patients with moderate/severe hypoxemic respiratory failure secondary to SARS-CoV-2 infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional oxygen therapy (COT) group (Active Comparator): Oxygen therapy will be delivered by conventional nasal cannula / prongs, venturi mask, or mask with reservoir, with flows between 3 and 15 liters / minute, to ensure SpO2 ≥ 92%.
  Interventions: Procedure: Conventional oxygen therapy
- High-flow nasal cannula (HFNC) group (Experimental): Breathing support with High-Flow oxygen therapy, flow will be initiated between 50 and 60 liters / minute. FiO2 60% to 100% with the objective of reaching SpO2 ≥ 92%. Adequate wetting of the system should be ensured according to the recommendations of the HFNC device manufacturer. FiO2 may be decreased gradually according to the patient's individual condition, trying to maintain SpO2 ≥ 92%.
  Interventions: Procedure: High flow nasal cannula

INTERVENTIONS:
Procedure: Conventional oxygen therapy — Oxygen therapy by conventional nasal cannula / prongs, venturi mask, or mask with reservoir
  Arms: Conventional oxygen therapy (COT) group
Procedure: High flow nasal cannula — Breathing support with High-flow nasal cannula
  Arms: High-flow nasal cannula (HFNC) group

SUMMARY:
This open label randomized controlled multicenter phase II trial will evaluate the clinical impact of the use of HFNC vs. conventional oxygen therapy in patients with moderate and severe hypoxemic acute respiratory failure secondary to SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure is a condition in which rapid-onset impairment in gas exchange between the lungs and the blood, lead to hypoxemia with or without hypercapnia. Usual management of this condition relies on oxygen supplementation throughout different respiratory support modalities (i.e., low flow oxygen devices, high-flow nasal cannulas, mechanical ventilation, ECMO, etc.) aiming to restore gas exchange and to support respiratory effort. In most cases, initial management of acute hypoxemic respiratory failure might be provided through low-flow oxygen systems, but more severe cases will require more advanced life-supporting strategies.

Respiratory compromise by SARS-CoV-2 infection widely varies between subjects. Thus, respiratory system elastance, intrapulmonary shunt, pulmonary perfusion/ventilation inequalities and lung weight can range between almost normal up to very high values. Consequently, modalities to provide initial support in acute severe hypoxemic respiratory failure in SARS-CoV-2 infection should not be limited to immediate invasive mechanical ventilation support as such respiratory support modalities should be adapted to individual requirements.

Unfortunately, similar values of initial PaO2/FiO2 ratios (especially when PaO2/FiO2 ratio is < 200) are not clearly related with more or less severe lung affectation, high or low respiratory system elastance patterns, high or low adaptive hypoxic vasoconstriction, and far beyond clinical signs, there are no widely available methods able to rapidly decide which patients would be more benefit from a relative "conservative" management or on the contrary, which patient would benefit from immediate invasive respiratory support.

Use of high-flow nasal cannulas (HFNC) in acute hypoxemic respiratory failure from different etiologies has rapidly increased during the last years. Certainly, randomized controlled trials suggest that HFNC might prevent intubation and the need for invasive mechanical ventilation in patients with moderate and severe hypoxemia. Nevertheless, impact of HFNC on mortality rates and other important clinical outcomes in this condition remains controversial.

Initial observational reports of patients with severe SARS-CoV-2 infection subjected to invasive mechanical ventilation showed a consistent and very high mortality. Indeed, some experts claimed for using such non-invasive respiratory support devices in patients with moderate or even high pulmonary shunt values arguing about possible harm induced by mechanical ventilation especially in patients with a relative normal respiratory system elastance. Nevertheless, others recommended against HFNC use because safety concerns for health care workers, which clearly limited its use at the initial phases of the pandemic. Thus, the impact and safety of using HFNC at very early stages of acute hypoxemic respiratory failure induced by severe SARS-CoV-2 infection remain to be elucidated. This is how the HiFlo-COVID trial propose to assess the impact HFNC vs. conventional oxygen therapy on the need for intubation / invasive mechanical ventilation support and the clinical status (at days-14 and -28) as assessed by a modified 7-point ordinal scale in patients with moderate / severe hypoxemic respiratory failure secondary to SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years.
* Emergency or ICU admission with suspected/confirmed SARS-CoV-2 infection.
* Moderate/severe acute respiratory failure:
* PaO2/FiO2 < 200.
* Use of accessory muscles.
* Breathing rate > 25 x minute.
* Have a progression < 6 hours since meeting the definition of moderate/severe acute respiratory failure secondary to suspected/confirmed SARS-CoV-2 infection.

Exclusion Criteria:

* Adults < 18 years.
* Indication for immediate orotracheal intubation.
* Pregnant woman / positive pregnancy test at the time of potential inclusion in the study.
* Chronic liver disease / liver cirrhosis Child-Pugh C.
* Confirmation of active bacterial or fungal infection.
* Uncontrolled HIV/AIDS disease (defined by presence of viral load > 200 copies/mL).
* Previous history of COPD Gold C - D.
* History of COPD requiring hospitalization - hospitalization / ICU in the last year.
* Known history of congestive heart failure NYHA III - IV.
* Left ventricular ejection fraction < 45% previously known.
* Highly suspected or confirmed cardiogenic pulmonary edema.
* Hypercapnic respiratory failure (PaCO2 > 55 mmHg).
* Central/peripheral demyelinating disorders due to medical history or high suspicion of these at the time of study eligibility.
* Patient who in the investigator's judgment suggests a progression to death is imminent and inevitable within the next 24 hours.
* Any serious medical condition or clinical laboratory test abnormality that, in the investigator's judgment, prevents safe patient participation and completion of the study.
* Participation in another clinical trial (except one related to SARS-CoV-2 - CRITERIA TO BE DISCUSSED BETWEEN GROUP OF RESEARCHES).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Intubation rate | 28 days
  Need for intubation / support with invasive mechanical ventilation.
Clinical recovery | 28 days
  Time to improvement of clinical status according to the 7-point ordinal scale.
  Modified 7-point ordinal scale:
  * An ordinal scale of 7 points where 1= Ambulatory/no limitation of activities and 7= Death. Low scores denote a better outcome and high scores denote a worse outcome.
  * Time to reduction in scale score will be measured (daily scale scoring).

SECONDARY OUTCOMES:
Proportion of patients with requirement of early mechanical ventilation. | 7 and 14 days
  Whether or not each patient required mechanical ventilation during the first 7 and 14 days after randomization will be assessed.
  Proportion of patients with early mechanical ventilation will be calculated for each group.
Mechanical ventilation-free days | 28 days
  Days off from mechanical ventilation
Renal replacement therapy-free days | 28 days
  Days off from renal replacement therapy
Length of ICU stay | 28 days
  Duration of stay in ICU
Length of hospital stay | 28 days
  Duration of hospital stay
All-cause day-28 mortality | 28 days
  Hospital mortality
Proportion of serious adverse events | 28 days
  Proportion of patients with serious adverse events during hospital stay
Proportion of bacterial - fungal infections | 28 days
  Proportion of bacterial - fungal infections during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A. Ospina Tascón, MDPhD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Derived] Ospina-Tascon GA, Calderon-Tapia LE, Garcia AF, Zarama V, Gomez-Alvarez F, Alvarez-Saa T, Pardo-Otalvaro S, Bautista-Rincon DF, Vargas MP, Aldana-Diaz JL, Marulanda A, Gutierrez A, Varon J, Gomez M, Ochoa ME, Escobar E, Umana M, Diez J, Tobon GJ, Albornoz LL, Celemin Florez CA, Ruiz GO, Caceres EL, Reyes LF, Damiani LP, Cavalcanti AB; HiFLo-Covid Investigators. Effect of High-Flow Oxygen Therapy vs Conventional Oxygen Therapy on Invasive Mechanical Ventilation and Clinical Recovery in Patients With Severe COVID-19: A Randomized Clinical Trial. JAMA. 2021 Dec 7;326(21):2161-2171. doi: 10.1001/jama.2021.20714. PMID 34874419